CLINICAL TRIAL: NCT01088685
Title: Feasibility Study to Evaluate the Safety and Performance of a Hydrogel Blister Patch Prototype for the Treatment of Foot Blisters
Brief Title: Hydrogel Blister Patch Prototype Treatment for Foot Blisters on the Heel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNKEDI0001
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Blister
MeSH Terms: conditions — Blister

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Blister Patch (Experimental): Experimental Hydrogel Blister patch
  Interventions: Device: Experimental Blister Patch
- Marketed Pflaster (Active Comparator): Scholls Blasen Pflaster
  Interventions: Device: Marketed Pflaster

INTERVENTIONS:
Device: Experimental Blister Patch — Experimental hydrogel blister patch to be applied as needed (at least every 2 days) consecutively until blister heals
  Other Names: No trade name available - not a marketed product
  Arms: Experimental Blister Patch
Device: Marketed Pflaster — Foot Blister Patch to be applied as needed (at least every 2 days) until blister heals
  Other Names: Scholls Blasen Pflaster
  Arms: Marketed Pflaster

SUMMARY:
Study to evaluate the safety and performance of a new blister patch intended to treat blisters on the heel of the foot.

DETAILED DESCRIPTION:
The study will require participation for up to 14 days of participation or less if the blister heals sooner, will recruit 100 subjects with fluid filled blisters on the heel of the foot that are intact and not broken. Some subjects will be asked to have their blisters photographed. All subjects will be required to have their blister unroofed (top layer of skin removed by the physician using sterile instruments). All subjects will receive study product, either test product or a marketed product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older;
* Individuals who are willing and able to provide informed consent
* Female subjects of child bearing potential must have a negative urine pregnancy test prior to application of the study products;
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to Visit 1 such as the ones listed below and agree to continue using this method during their participation in the study; Note that abstinence is not an approved method of birth control.

  * Postmenopausal or amenorrheic for one year
  * Surgically sterile (hysterectomy, tubal ligation, or oophorectomy)
  * Use of an effective method of birth control (e.g. prescription oral contraceptives, contraceptive implants or injections, intrauterine device, diaphragm, cervical cap or condoms with spermicide)
* Individuals exhibit a blister on the heel that is determined by the investigator to be no more than 72 hours old and in stage 2
* Subject is willing to have blister unroofed (top layer of blister removed) by the investigator
* Subject is willing and able to follow the study directions, to participate in the study, and to return for all specified visits

Exclusion Criteria:

* Pregnant, planning a pregnancy or actively nursing
* Exhibits a foot blister on the heel that exceeds 1125mm2 or would otherwise not be covered by the hydrogel portion of the study product
* Unstable or uncontrolled medical conditions that could require intensive treatment during the course of the study
* Individuals with autoimmune disorders including, but not limited to, lupus erythematosus, rheumatoid arthritis, or HIV/AIDS
* Currently participating in or, within the past 30 days have participated in another clinical study using an investigational drug or device
* Employees of the site, or friends/relatives of employees that would have access to study information
* Diabetic, type I or type II
* Treatment for any type of cancer within the last 2 years or history of skin cancer
* Damaged skin in or around test sites, which include sunburn, extremely deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, acne, and disfiguration of the test site
* History of clinically determined allergic reaction or irritation to any of the test product ingredients
* History of or known allergy to iodine
* Currently taking or expected to take any of the following during the course of the study: amphetamines, benzodiazepines, cocaine, marijuana, methaqualone, methadone, opiates, propoxyphene, barbiturates, and phencyclidine
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Investigator Assessment | at subject's last visit, within 14 days of start
  Global assessment of the product by the investigator at the subject's last visit.

SECONDARY OUTCOMES:
Subject Assessment | at subject's last visit, within 14 days of start
  Global assessment of the product by the subject at the subject's last visit.
Time to Heal | Baseline to subject's last visit, within 14 days of start
  Record of the time it took for the blister to heal within the 14-day study period.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, PhD, Study Director — J&J Consumer and Personal Products Worldwide
Locations (1):
- SCIderm GmbH, Hamburg, Germany